CLINICAL TRIAL: NCT03743597
Title: SOCKNLEG Leg Compression Stocking Kit: Physical Properties: Static Stiffness Index - Venous Ejection Fraction An Open Monocentric Randomized Controlled Cross-over Trial
Brief Title: SOCKNLEG Compression Stocking Kit: Physical Properties
Acronym: SOCKNLEGLCA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SL1726
Record Dates: First submitted 2018-11-13; First posted 2018-11-16 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Venous Insufficiency of Leg

STUDY DESIGN:
Intervention Model Description: A computer generated list will allocate each participant to either one of the stockings, the innovative SOCKNLEG, or the standard Sigvaris COTTON stocking. In each participant the examinations will be conducted with both stockings.
  The allocated group defines with which stocking the examinations will be conducted first.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SOCKNLEG (Experimental): Group of participant who will conduct the examinations first with the SOCKNLEG compression stockings.
  All examinations will be conducted in all participants and with both stockings one after the other.
  Interventions: Device: SOCKNLEG; Device: Sigvaris COTTON
- Sigvaris COTTON (Active Comparator): Group of participant who will conduct the examinations first with the Sigvaris COTTON compression stockings.
  All examinations will be conducted in all participants and with both stockings one after the other.
  Interventions: Device: SOCKNLEG; Device: Sigvaris COTTON

INTERVENTIONS:
Device: SOCKNLEG — Innovative multilayer leg compression stocking, compression strength CEN compression class II (European Compression Strength) with compression at the ankle of 23-32mmhg, product composition understocking (polyamide, cotton, spandex), overstocking (polyamide, spandex)
  In each participant all examinations will be performed with both study stockings, one after the other
Device: Sigvaris COTTON — Standard single leg compression stocking, compression strength CEN compression class II (European Compression Strength) with compression at the ankle of 23-32mmhg, product composition one stocking (polyamide, spandex, cotton)
  In each participant all examinations will be performed with both study stockings, one after the other

SUMMARY:
This study evaluates physical properties of a innovative leg compression stocking compared to a standard compression stocking of the same compression strength in patients with chronic venous insufficiency clinical stadium C3 and above, according to the CEAP classification for chronic venous insufficiency.

The physical properties can be measured through a series of measurements. The hypothesis is that the innovative compression stocking, although changed in design to be more easily donned, will perform as good as the standard compression stocking.

In each participant the examinations will be conducted with both stockings. A computer generated list will allocate each participant to either one of the stockings, with which the examinations will be conducted first.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Male or post-menopausal women over the age of 65
* Diagnosed chronic venous insufficiency stage C3-C6 (according to CEAP classification)
* Indication of a compression therapy by medical compression stocking

Exclusion Criteria:

* Peripheral artery disease (PAD) or calcinosis (Ankle-Brachial-Index <0.8 or >1.3
* Suspected polyneuropathy with ≤4 sensible test areas measured with the Semmes- Weinstein-Monofilament-Test
* Advanced heart insufficiency (NYHA III-IV)
* Contraindications to compression therapy
* Known allergies to any components of the stocking material
* Inability to follow the procedures of the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2018-11-19 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Static Stiffness Index (SSI) values of both stockings in mmHg measured at point cB1 on the leg | 1 day, during study visit
  The SSI is a substraction of the Interface Pressures measured with a pressure probe on the leg of the study participant in standing and in supine position while wearing a compression stocking. The point cB1 is a thereby a standard measuring point at the distal insertion of the gastrocnemius muscle of the leg.

SECONDARY OUTCOMES:
Static Stiffness Index (SSI) values of both stocking in mmHg measured at point cC on the leg | 1 day, during study visit
  Comparing the SSI at point cC of both stockings with each other and with the standard SSI values at point cB1. The point cC is a new measuring point at the largest circumference of the calf.
Dynamic Stiffness Index (DSI) values of both stockings in mmHg | 1 day, during study visit
  The DSI is a substraction of the Interface Pressures measured at each point (cC and cB1) on the leg during wiping of the foot while wearing a compression stocking. Measuring instruments are again the pressure probes.
Venous ejection fraction (VEF) of both stockings in % | 1 day, during study visit
  Non-invasive measurement of the venous filling volumes of the leg with a strain gauge plethysmography the Angioflow2 (Microlabitalia, Padua, Italy).
Interface Pressures at point cB on the leg in mmHg | 1 day, during study visit
  The point cB is the point of the smallest circumference of the leg and is the standard measuring point for compression strength of a leg compression stocking. Measured with a pressure probe on the leg of the study participant under the compression stocking.

CONTACTS AND LOCATIONS:
Overall Officials: Juerg Hafner, M.D. Prof., Principal Investigator — Department of Dermatology, University Hospital Zurich, Zurich, Switzerland
Locations (1):
- Department of Dermatology, University Hospital of Zurich, Switzerland, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No